CLINICAL TRIAL: NCT06005246
Title: Munich Cohort Study With Biobank for Children, Adolescents, and Young Adults With Post-infection ME/CFS (MUC-CFS)
Brief Title: Munich ME/CFS Cohort Study
Acronym: MUC-CFS
Status: Recruiting | Type: Observational
Sponsor: Technical University of Munich (Other)
Collaborators: Helmholtz Munich, Munich (Unknown); German Cancer Research Center (Other); Charité University Hospital, Berlin, Germany (Unknown)
Responsible Party: Sponsor
Other Study IDs: MUC-CFS
Record Dates: First submitted 2023-07-24; First posted 2023-08-22 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-07

CONDITIONS: Myalgic Encephalomyelitis/Chronic Fatigue Syndrome (ME/CFS) (ICD-10 G93.3)
Keywords: ME/CFS; CFS/ME; SEID; myalgic encephalomyelitis; chronic fatigue syndrome; infectious mononucleosis; systemic exertion intolerance disease; Epstein-Barr virus; post-COVID-19-syndrome; post-COVID-19 condition; long COVID; post-acute sequelae of COVID-19
MeSH Terms: conditions — Fatigue Syndrome, Chronic; Infectious Mononucleosis; Epstein-Barr Virus Infections; Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Munich cohort study MUC-CFS aims at the characterization and long-term follow-up of myalgic encephalitis/chronic fatigue syndrome (ME/CFS) in young people aged up to 25 years, as well as at the identification of pathomechanisms, biomarkers, and targets for future treatment approaches.

DETAILED DESCRIPTION:
ME/CFS is a complex, chronic neurological disorder with an estimated pre-pandemic prevalence of about 0.3%, affecting more people than multiple sclerosis (MS) worldwide. The number of cases was reported to increase due to long-term sequelae of COVID-19 (post-COVID condition). ME/CFS mainly affects young females aged 15-40 years but can occur in males and children. 25% are mildly, 50% moderately, and 25% severely affected.

Patients with ME/CFS suffer from fatigue, exertion intolerance with post-exertional malaise (PEM), cognitive impairment, pain, sleep disturbances, autonomic, and neuroendocrine manifestations, and flu-like symptoms. ME/CFS accounts for many cases of long-term school or work absences, with subsequent high social and economic burdens. The health-related quality of life is lower than in other severe chronic diseases.

Most ME/CFS cases are triggered by an infection-like event (so-called post-infection ME/CFS). Prominent triggers of ME/CFS include Epstein-Barr virus-associated infectious mononucleosis (EBV-IM) and coronavirus disease 2019 (COVID-19). Moreover, cases following other infectious diseases (e.g., other COVID, Influenza, Dengue fever, Ebola) are well documented.

Possible mechanisms contributing to the pathogenesis of ME/CFS include reactivation of latent viral infections, chronic inflammation, and autoimmunity, resulting in metabolic, neurological, and vascular dysregulation. However, no biomarker or causative treatment for ME/CFS has been established yet.

ME/CFS (ICD10 G93.3) affords appropriate differential diagnostics and is defined by clinical criteria. The criteria most commonly used are the criteria for "systemic exertion intolerance disease (SEID) defined by the former Institute of Medicine (IOM) and the Canadian Consensus Criteria (CCC). Adapted pediatric criteria have been suggested by the groups of P.C. Rowe and L.A. Jason in the US.

ME/CFS treatment includes comprehensive patient education regarding self-management strategies (e.g., pacing, relaxation strategies, sleep hygiene) as well as pharmaceutical and non-pharmaceutical approaches to palliate symptoms such as pain, sleep disorder, or orthostatic intolerance. Appropriate psychosocial support for patients and their families is essential. Follow-up studies indicated a better prognosis in children compared to adults.

The MUC-CFS cohort study is recruiting patients from the MRI Chronic Fatigue Center for Young People (MCFC) at the Technical University of Munich (TUM) and the Munich Municipal Hospital (MüK) in Munich, Germany. The MCFC closely cooperates with the Charité Fatigue Center (CFC) in Berlin, Germany, and has long-standing expertise in ME/CFS care and research.

The MUC-CFS cohort study aims to collect comprehensive clinical data regarding medical history, clinical and laboratory phenotypes, the trajectory of individual diseases, health-related quality of life, education, and social participation. Clinical data are derived from complex initial investigations at in- or out-patient visits as well as from following telephone calls and from various questionnaires. Biosampling (blood, urine, and/or mouthwashes) takes place at any personal visit for later cell-analytical, molecular, and/or biochemical analyses by our study group.

ELIGIBILITY:
Inclusion Criteria:

* Written consent of the patient (or legal guardian for patients aged < 18 years).
* Age 0 - 25 (including)
* Documented or probable acute infectious disease at the onset of ME/CFS symptoms
* Diagnosis of ME/CFS according to the IOM criteria, the CCC, the diagnostic worksheet published by P.C. Rowe et al. (2017), or the pediatric case definition published by L.A. Jason et al. (2006).

Exclusion Criteria:

• drug/medication abuse, major surgery within the last six months, presence of organ failure, post-stroke/craniocerebral trauma with cognitive deficits, post-intensive care syndrome, syphilis, Lyme disease, AIDS, hepatitis B/C, multiple sclerosis, systemic lupus erythematosus, Sjörgren's syndrome, malignancy, major depression or other severe psychiatric illness, primary sleep disorder, severe endocrine disease (e.g., hypopituitarism, adrenal insufficiency), and other conditions that might explain ME/CFS symptoms.

Max Age: 25 Years | Sex: All
Age Groups: Child, Adult
Study Population: The number of study participants will not be limited.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-01-22 (Actual); Primary Completion 2024-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Extensive Phenotyping of ME/CFS Patients | 5 years
  Extensive phenotyping of children, adolescent, and young adult patients with post-infectious ME/CFS (e.g., age, gender, medical history, daily function, health-related quality of life, severity and frequency of symptoms, disease trajectory over time)

SECONDARY OUTCOMES:
Risk factors | 5 years
  Identification of risk factors for protracted courses without (partial) remission (e.g., age at symptom onset, sex, sociodemographic variables, medical history, medication, daily function at symptom onset, severity and frequency of symptoms at symptom onset, laboratory values, EBV serology, EBV DNA load).
Biomarkers | 5 years
  Identification of diagnostic biomarkers, i.e., a single and/or a combination of which, indicative of post-infectious ME/CFS (e.g., inflammatory markers, autoantibodies, EBV serology, EBV DNA load).

CONTACTS AND LOCATIONS:
Overall Officials: Uta Behrends, Prof. Dr., Principal Investigator — München Klinik Schwabing
Locations (1):
- MRI Chronic Fatigue Center for Young People (MCFC), Children's hospital, Technical University of Munich (TUM) and Munic Municipal Hospital (MüK), Munich, Bavaria, Germany

REFERENCES:
- [Background] Pricoco R, Meidel P, Hofberger T, Zietemann H, Mueller Y, Wiehler K, Michel K, Paulick J, Leone A, Haegele M, Mayer-Huber S, Gerrer K, Mittelstrass K, Scheibenbogen C, Renz-Polster H, Mihatsch L, Behrends U. One-year follow-up of young people with ME/CFS following infectious mononucleosis by Epstein-Barr virus. Front Pediatr. 2024 Jan 18;11:1266738. doi: 10.3389/fped.2023.1266738. eCollection 2023. PMID 38304441
- See also: Homepage of the MRI Chronic Fatigue Center for Young People (MCFC) — https://www.mri.tum.de/chronische-fatigue-centrum-fuer-junge-menschen-mcfc